CLINICAL TRIAL: NCT02092831
Title: A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE EFFECT OF FORMULATION AND TABLET HARDNESS ON THE RELATIVE BIOAVAILABILITY OF PICTILISIB (GDC-0941) IN HEALTHY SUBJECTS
Brief Title: A Study of the Effect of Formulation and Tablet Hardness on the Bioavailability of Pictilisib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP29284
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

ARMS (4):
- Crossover sequence 1 (Experimental)
  Interventions: Drug: GDC-0941
- Crossover sequence 2 (Experimental)
  Interventions: Drug: GDC-0941
- Crossover sequence 3 (Experimental)
  Interventions: Drug: GDC-0941
- Crossover sequence 4 (Experimental)
  Interventions: Drug: GDC-0941

INTERVENTIONS:
Drug: GDC-0941 — Single dose market image tablet of hardness 1
Drug: GDC-0941 — Single dose market image tablet of hardness 2
Drug: GDC-0941 — Single dose market image tablet of hardness 3
Drug: GDC-0941 — Single dose Phase 2 tablet formulation

SUMMARY:
This Phase 1, open-label, randomized, 4-period crossover study is designed to determine the relative bioavailability of GDC-0941 administered as a single dose of the market image formulation at 3 different hardnesses (hardness 1, 2, and 3) and as a single dose of the Phase 2 formulation to healthy male and female volunteers. Participants will be randomly assigned to 4 possible treatment sequences, each comprising 4 periods (1 per formulation), and GDC-0941 will be administered based on the assigned sequence. The study is expected to last 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 55 years of age, inclusive,
* Body mass index (BMI) between 18.5 to 32 kg/m2, inclusive,
* Healthy, as determined by no clinically significant findings from medical history, ECG, and vital signs, and who are able to swallow and tolerate a tethered Heidelberg pH Capsule and have gastric pH measurements taken

Exclusion Criteria:

* Any medical condition or history of such condition that may, in the opinion of the investigator, contraindicate participation in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of plasma GDC-0941 | 25 Days
Maximum plasma concentration (Cmax) of GDC-0941 | 25 Days
Relative bioavailability (Frel) according to the model independent approach | 25 days

SECONDARY OUTCOMES:
Incidence of adverse events | 25 days
Electrocardiogram (ECG) | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madison, Wisconsin, United States